CLINICAL TRIAL: NCT00640263
Title: A Randomised Controlled Trial Comparing the Efficacy of Infant Peri-exposure Prophylaxis With Lopinavir/Ritonavir (LPV/r) Versus Lamivudine to Prevent HIV-1 Transmission by Breastfeeding
Brief Title: Comparison of Efficacy and Safety of Infant Peri-exposure Prophylaxis With Lopinavir/Ritonavir Versus Lamivudine to Prevent HIV-1 Transmission by Breastfeeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); The Research Council of Norway (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government); Université Montpellier (Other); University of Bergen (Other)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANRS 12174 PROMISE-PEP; EDCTP : RCN 183600
Record Dates: First submitted 2008-01-15; First posted 2008-03-21 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Breastfeeding; Prevention; lamivudine; lopinavir/ritonavir
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Lopinavir; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): infant peri-exposure prophylaxis with lopinavir/ritonavir
  Interventions: Drug: lopinavir/ritonavir (LPV/r)
- 2 (Active Comparator): infant peri-exposure prophylaxis with lamivudine
  Interventions: Drug: Lamivudine (3TC)

INTERVENTIONS:
Drug: lopinavir/ritonavir (LPV/r) — Oral liquid formulation lopinavir/ritonavir(80 mg lopinavir + 20 mg ritonavir/mL); Dosing : 40/10mg twice daily if infant weight is between 2 to 4 kg and 80/20mg twice daily if infant weight is above 4kg The lopinavir/ritonavir will be given to the baby from Day 7 postnatal until 4 weeks after the cessation of breastfeeding. During the treatment period, dosing will be adapted according to the infant weight.
  Arms: 1
Drug: Lamivudine (3TC) — Oral liquid solution lamivudine(10 mg/mL). Dosing : 7,5 mg twice daily if if infant weight is between 2 to 4 kg ; 25 mg twice daily if infant weight is between 4 to 8 kg ; 50 mg twice daily if infant weight is above 8kg.
  The lamivudine will be given to the baby from Day 7 postnatal until 4 weeks after the cessation of breastfeeding. During the treatment period, dosing will be adapted according to the infant weight.
  Arms: 2

SUMMARY:
The ANRS 12174 study is a clinical trial that will compare the efficacy and safety of prolonged infant peri-exposure prophylaxis (PEP) with Lopinavir/Ritonavir (LPV/r) versus Lamivudine to prevent HIV-1 transmission through breast milk in children born to HIV-1-infected mothers not eligible for HAART and having benefited from perinatal antiretroviral (ART) regimens. The study will recruit 1500 mother-infant pairs in 4 African countries.

Study design:

PROMISE PEP is a multinational, randomised double-blind controlled clinical trial.

Intervention:

Infants will be randomised to receive LPV/r or 3TC twice daily from day seven (± 2 days) after birth until 4 weeks after cessation of breastfeeding (BF). We will recommend exclusive BF (EBF) up till including the 26th week of life followed by a relatively rapid (maximum of 8 weeks) cessation period. The maximum duration of PEP will thereby be 38 weeks.

Primary objective:

To compare the efficacy of infant LPV/r (40/10mg twice daily if 2-4kg and 80/20mg twice daily if >4kg) vs. Lamivudine 7,5mg twice daily if 2-4kg, 25mg twice daily if 4-8kg and 50mg twice daily if >8kg) from day 7 until 4 weeks after cessation of BF (maximum duration of prophylaxis: 50 weeks for a maximum duration of breastfeeding of 46 weeks) to prevent postnatal HIV-1 acquisition between 7 days and 50 weeks of age.

Secondary objectives:

* To assess the safety of long-term infant prophylaxis with LPV/r versus Lamivudine (including resistance, adverse events and growth) until 50 weeks.
* HIV-1-free survival until 50 weeks
* To build clinical trials capacity at the four study sites.

Main endpoint:

Acquisition of HIV-1 (as assessed by HIV-1 DNA PCR) between day 7 and 50 weeks of age

Study population:

HIV-uninfected infants at day 7 (± 2 days) born to HIV-1 infected mothers not eligible for HAART who choose to breastfeed their infants and who have benefited from the national prevention of mother to child transmission (PMTCT) program during pregnancy and delivery. The study will recruit 1500 mother-infant pairs in Burkina Faso, South Africa, Uganda and Zambia.

Study duration:

Infants will be followed up for 50 weeks and the total study duration is five years.

Expected outcome:

This study will inform on the relative advantages (efficacy) and drawbacks of two interventions to support HIV-1-infected women not eligible for HAART to safely breastfeed their babies. If found to be safe and efficacious, the regimens would avoid the existing contradiction between optimal infant feeding and the prevention of MTCT through breast milk. Clinical trial capacity development will improve the future quality of trials conducted in these countries.

ELIGIBILITY:
Inclusion Criteria: A baby will be included if she/he:

* is a singleton
* is breastfed at day 7 by her/his mother and her/his mother intends to continue breastfeeding for at least 6 months
* has a post-partum blood sample with a negative HIV-1 DNA PCR test result at day 7 (+/- 2 days)
* has received ART as part of PMTCT

and if the mother:

* has reached the local legal age for participating in medical research studies
* is shown to be HIV-1 infected (with or without HIV-2 infection) and is not eligible for HAART or is not taking HAART
* has received a perinatal antiretroviral prophylaxis during pregnancy and delivery,
* has a CD4 count above the threshold of HAART initiation in pregnant women according to the national recommendation in each site (minimum 230 cells/µL),
* resides within the study area and is not intending to move out of the area in the next year
* gives assent for the infant to participate and gives consent to participate

Exclusion Criteria:

* S/he presents clinical symptoms and/or biological abnormalities equal to or greater than grade II of the ANRS classification for adverse event on the day of enrolment
* S/he presents with serious congenital malformation(s)
* Her/his birth weight is lower than 2.0 kg
* Her/his antiretroviral prophylaxis is extending beyond day 7
* The mother has participated in the trial for a previous pregnancy
* S/he and her/his mother are participating in another clinical trial on the day of enrolment

Ages: 5 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Acquisition of HIV-1 (as determined by HIV-1 DNA PCR) | between day 7 and 50 weeks of age

SECONDARY OUTCOMES:
HIV-1 free survival | at 50 weeks of age
HIV-1 free survival | at one year of age
safety of long-term prophylaxis | until 50 weeks of age
safety of long-term prophylaxis | until one year of age

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Vande Perre, MD, PhD, Study Chair — University of Montpellier, France; Thorkild Tylleskär, MD, PhD, Study Chair — Centre For International Health; Nicolas Meda, MD, PhD, Principal Investigator — University of Ouagadougou, Burkina Faso; James K Tumwine, MD, PhD, Principal Investigator — Dept of Paediatrics and Child Health, Makerere University, Uganda; Chipepo Kankasa, MD, Principal Investigator — Dept of Paediatrics and Child Health, School of Medicine, University of Zambia; Justus Hofmeyer, MD, Principal Investigator — East London Hospital Complex; Eva-Charlotte Ekström, PhD, Principal Investigator — Uppsala University, Uppsala, Sweden; Stephane Blanche, MD, PhD, Principal Investigator — Hôpital Necker Enfants Malades, Université Paris V (EA 3620)
Locations (4):
- Université de Ouagadougou, Ouagadougou, Burkina Faso
- East London Hospital Complex, East London, South Africa
- Dept of Paediatrics and Child Health, Makerere University, Kampala, Uganda
- Dept of Paediatrics and Child Health, School of Medicine, University of Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Kourtis AP, Jamieson DJ, de Vincenzi I, Taylor A, Thigpen MC, Dao H, Farley T, Fowler MG. Prevention of human immunodeficiency virus-1 transmission to the infant through breastfeeding: new developments. Am J Obstet Gynecol. 2007 Sep;197(3 Suppl):S113-22. doi: 10.1016/j.ajog.2007.03.003. PMID 17825642
- [Derived] Birungi N, Fadnes LT, Engebretsen IMS, Tumwine JK, Astrom AN; for ANRS 12174 AND 12341 study groups. Antiretroviral treatment and its impact on oral health outcomes in 5 to 7 year old Ugandan children: A 6 year follow-up visit from the ANRS 12174 randomized trial. Medicine (Baltimore). 2020 Sep 25;99(39):e22352. doi: 10.1097/MD.0000000000022352. PMID 32991450
- [Derived] Birungi N, Fadnes LT, Engebretsen IMS, Lie SA, Tumwine JK, Astrom AN; ANRS 12174 and 12341 study groups. Caries experience and oral health related quality of life in a cohort of Ugandan HIV-1 exposed uninfected children compared with a matched cohort of HIV unexposed uninfected children. BMC Public Health. 2020 Mar 30;20(1):423. doi: 10.1186/s12889-020-08564-1. PMID 32228542
- [Derived] Montoya-Ferrer A, Sanosyan A, Fayd'herbe de Maudave A, Pisoni A, Bollore K, Moles JP, Peries M, Tylleskar T, Tumwine JK, Ndeezi G, Gorgolas M, Nagot N, van de Perre P, Tuaillon E. Clinical and Biological Factors Associated With Early Epstein-Barr Virus Infection in Human Immunodeficiency Virus-Exposed Uninfected Infants in Eastern Uganda. Clin Infect Dis. 2021 Mar 15;72(6):1026-1032. doi: 10.1093/cid/ciaa161. PMID 32067040
- [Derived] Birungi N, Fadnes LT, Engebretsen IMS, Lie SA, Tumwine JK, Astrom AN; ANRS 12174 and 12341 study groups. Association of maternal HIV-1 severity with dental caries: an observational study of uninfected 5- to 7-yr-old children of HIV-1-infected mothers without severe immune suppression. Eur J Oral Sci. 2020 Feb;128(1):46-54. doi: 10.1111/eos.12669. Epub 2020 Jan 29. PMID 31994250
- [Derived] Kariyawasam D, Peries M, Foissac F, Eymard-Duvernay S, Tylleskar T, Singata-Madliki M, Kankasa C, Meda N, Tumwine J, Mwiya M, Engebretsen I, Fluck CE, Hartmann MF, Wudy SA, Hirt D, Treluyer JM, Moles JP, Blanche S, Van De Perre P, Polak M, Nagot N; ANRS 12174 Trial Group. Lopinavir-Ritonavir Impairs Adrenal Function in Infants. Clin Infect Dis. 2020 Aug 14;71(4):1030-1039. doi: 10.1093/cid/ciz888. PMID 31633158
- [Derived] Blanche S, Tylleskar T, Peries M, Kankasa C, Engebretsen I, Meda N, Tumwine JK, Singata-Madliki M, Mwiya M, Van de Perre P, Nagot N; ANRS 12174 Trial Group. Growth in HIV-1-exposed but uninfected infants treated with lopinavir-ritonavir versus lamivudine: a secondary analysis of the ANRS 12174 trial. Lancet HIV. 2019 May;6(5):e307-e314. doi: 10.1016/S2352-3018(18)30361-8. Epub 2019 Feb 24. PMID 30814028
- [Derived] Some EN, Engebretsen IMS, Nagot N, Meda N, Lombard C, Vallo R, Peries M, Kankasa C, Tumwine JK, Hofmeyr GJ, Singata M, Harper K, Van De Perre P, Tylleskar T; ANRS 12174 Trial Group. Breastfeeding patterns and its determinants among mothers living with Human Immuno-deficiency Virus -1 in four African countries participating in the ANRS 12174 trial. Int Breastfeed J. 2017 May 2;12:22. doi: 10.1186/s13006-017-0112-2. eCollection 2016. PMID 28469697
- [Derived] Foissac F, Blume J, Treluyer JM, Tylleskar T, Kankasa C, Meda N, Tumwine JK, Singata-Madliki M, Harper K, Illamola SM, Bouazza N, Nagot N, Van de Perre P, Blanche S, Hirt D. Are Prophylactic and Therapeutic Target Concentrations Different?: the Case of Lopinavir-Ritonavir or Lamivudine Administered to Infants for Prevention of Mother-to-Child HIV-1 Transmission during Breastfeeding. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01869-16. doi: 10.1128/AAC.01869-16. Print 2017 Feb. PMID 27895016
- [Derived] Nagot N, Kankasa C, Tumwine JK, Meda N, Hofmeyr GJ, Vallo R, Mwiya M, Kwagala M, Traore H, Sunday A, Singata M, Siuluta C, Some E, Rutagwera D, Neboua D, Ndeezi G, Jackson D, Marechal V, Neveu D, Engebretsen IMS, Lombard C, Blanche S, Sommerfelt H, Rekacewicz C, Tylleskar T, Van de Perre P; ANRS 12174 Trial Group. Extended pre-exposure prophylaxis with lopinavir-ritonavir versus lamivudine to prevent HIV-1 transmission through breastfeeding up to 50 weeks in infants in Africa (ANRS 12174): a randomised controlled trial. Lancet. 2016 Feb 6;387(10018):566-573. doi: 10.1016/S0140-6736(15)00984-8. Epub 2015 Nov 19. PMID 26603917
- [Derived] Nagot N, Kankasa C, Meda N, Hofmeyr J, Nikodem C, Tumwine JK, Karamagi C, Sommerfelt H, Neveu D, Tylleskar T, Van de Perre P; PROMISE-PEP group. Lopinavir/Ritonavir versus Lamivudine peri-exposure prophylaxis to prevent HIV-1 transmission by breastfeeding: the PROMISE-PEP trial Protocol ANRS 12174. BMC Infect Dis. 2012 Oct 6;12:246. doi: 10.1186/1471-2334-12-246. PMID 23039034